CLINICAL TRIAL: NCT04856371
Title: A Multicenter, Open-label, Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CYH33 in Combination With Endocrine Therapy With or Without Palbociclib in Patients With PIK3CA Mutant, HR+, HER2- Advanced Breast Cancer
Brief Title: Study of CYH33 in Combination With Endocrine Therapy With or Without Palbociclib in Patients With HR+, HER2- Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYH33-G103
Record Dates: First submitted 2021-04-11; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Advanced Breast Cancer
Keywords: PIK3CA Mutant; Advanced Breast Cancer
MeSH Terms: interventions — CYH33; Fulvestrant; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CYH33 + fulvestrant (Experimental): Participants will receive CYH33 in combination with a standard fixed dose of fulvestrant 500 mg.
  Interventions: Drug: CYH33; Drug: Fulvestrant
- CYH33 + fulvestrant + palbociclib (Experimental): Participants will receive CYH33 in combination with standard fixed dose of fulvestrant (500 mg) and palbociclib (125 mg).
  Interventions: Drug: CYH33; Drug: Fulvestrant; Drug: Palbociclib
- CYH33 + letrozole + palbociclib (Experimental): Participants will receive CYH33 in combination with standard fixed dose of letrozole (2.5 mg) and palbociclib (125 mg)
  Interventions: Drug: CYH33; Drug: Letrozole; Drug: Palbociclib

INTERVENTIONS:
Drug: CYH33 — Participants will receive oral CYH33 once daily on Days 1-28 of each 28-day cycle.
Drug: Fulvestrant — Participants will receive fulvestrant 500 mg, administered intramuscularly on Days 1, 15 on Cycle 1 (28-day cycle) and Day 1 at each 28-day cycle thereafter.
  Arms: CYH33 + fulvestrant; CYH33 + fulvestrant + palbociclib
Drug: Letrozole — Participants will receive oral letrozole once daily continuous on Day 1-28 of each cycle.
  Arms: CYH33 + letrozole + palbociclib
Drug: Palbociclib — Participants will receive palbociclib once daily continuous on Day 1-21 of each 28-day cycle.
  Arms: CYH33 + fulvestrant + palbociclib; CYH33 + letrozole + palbociclib

SUMMARY:
This is a multicenter, open-label, phase Ib study designed to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of CYH33 administered orally in combination with standard-of-care ET ± CDK4/6 inhibitor therapies for the treatment of locally advanced, recurrent or metastatic hormone-receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) breast cancer. Patients will be enrolled in two stages, including dose exploration phase (Stage 1) and dose expansion phase (Stage 2) of each cohort.

ELIGIBILITY:
Main Inclusion Criteria:

1. Provide informed consent voluntarily.
2. Male and female patients ≥ 18 years of age.
3. Patient must have a histologically or cytologically documented locally advanced, recurrent or metastatic breast cancer.
4. In case of women, both premenopausal and postmenopausal patients can be enrolled in the study.
5. Confirmed diagnosis of HR+, HER2- breast cancer.
6. For Stage 1 dose exploration phase, patients with or without PIK3CA mutation may be enrolled; For Stage 2 dose expansion phase, patients with PIK3CA mutations are required.
7. Patient must have evidence of disease radiological progression after previous endocrine therapy, or other systemic therapy.
8. Patient has measurable disease per RECIST v1.1.
9. ECOG ≤ 1.
10. Patient must have adequate organ and bone marrow function.

Main Exclusion Criteria:

1. Previously received any anticancer therapy within 28 days or 5 times of half-lives prior to the first dose of the study treatment.
2. Previously received treatment with any PI3Kα inhibitor, AKT inhibitor, or mTOR inhibitor.
3. Radical radiation therapy within 4 weeks prior to the first dose of the study treatment.
4. Patient with an established diagnosis of diabetes mellitus.
5. Any other concurrent disease with potential risk of insulin resistance or current use of medication with potential risk of insulin resistance.
6. Patient with clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 28 days
  Incidence rate of DLT in the first cycle (of 28 days).

SECONDARY OUTCOMES:
Safety and tolerability | 30 months
  Type, incidence, duration, severity and seriousness of adverse events (AEs).
Preliminary efficacy-ORR | 30 months
  Tumor objective response rate (ORR) assessed by RECIST v1.1
Preliminary efficacy-CBR | 30 months
  Clinical benefit rate (CBR) assessed by RECIST v1.1
Preliminary efficacy-PFS | 30 months
  Progression Free Survival (PFS) assessed by RECIST v1.1
Pharmacokinetic measures - AUC | 20 months
  Measure the variation of concentration in blood plasma as a function of time
Pharmacokinetic measures - C trough | 20 months
  Measure the minimum (trough) plasma concentration
Pharmacokinetic measures - Cmax | 20 months
  Measure the maximum (peak) plasma concentration
Pharmacokinetic measures - Tmax | 20 months
  Measure of time to reach maximum (peak) plasma concentration
Pharmacokinetic measures - CL/F | 20 months
  Measure apparent total clearance(s) from plasma after administration
Pharmacokinetic measures - Vz/F | 20 months
  Measure apparent volume of distribution during terminal phase
Assess downstream effects of PI3K pathway inhibition on blood glucose | 20 months
  Pre- and post-treatment of blood glucose
Assess downstream effects of PI3K pathway inhibition on C peptide | 20 months
  Pre- and post-treatment of C peptide
Assess the changes of biomarker-PIK3CA | 20 months
  Pre- and post-treatment PIK3CA changes in ctDNA samples.
Assess the changes of biomarker-PTEN | 20 months
  Pre- and post-treatment PTEN changes in ctDNA samples.
Assess the changes of biomarker-KRAS | 20 months
  Pre- and post-treatment KRAS changes in ctDNA samples.